CLINICAL TRIAL: NCT03566472
Title: The Current Situation and Influence Factors of Blood Glucose Control in Patients With Type 2 Diabetes Treated With Glargine in China
Brief Title: The Blood Glucose Control in Patients With Type 2 Diabetes Treated With Glargine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20170904-05
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2018-06

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Continuous Glucose Monitoring System — Continuous Glucose Monitoring System for 72 hours

SUMMARY:
Glargine is commonly used in insulin supplemental therapy in patients with type 2 diabetes(T2D) at present. This study aims to investigate the current status of blood glucose control in patients with T2D treated with glargine. Glycated hemoglobin(HbA1c) will be tested in these patients to assess the blood glucose control and Continuous Glucose Monitoring System (CGMS) will be used to investigate the glucose variability. Islet function, duration of diabetes, complications, exercise, insulin dose, oral medication regimen and insulin antibodies will be recorded in detail. This study will analysis the association between these clinical characteristics and blood glucose control.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM, which was defined bypublished Criteria of World Health Organization in 1999;
2. Patients were using glargine with or without oral hypoglycemic drugs and having a stable dose of glargine for more than 2 month would be recruited into this study;
3. Patients had relatively constant diet and exercise in 2 month before the study;
4. Fasting blood glucose was between 6.1 and 16mmolL, and postprandial (or random) blood glucose <22.2mmol/L.

Exclusion Criteria:

1. Patients with severe cardiovascular diseases, such as stroke, transient ischemic attack, myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous coronary intervention, and heart failure;
2. Patients with severe infectious diseases;
3. Patients with acute complications of diabetes on admission, such as diabetic ketoacidosis, diabetic hyperosmolar nonketotic coma, and lactic acidosis;
4. Patients with history of psychiatric disorders and were unsuitable to use CGMS;
5. Any other situations that made patients unsuitable to participate in the study, such as alcoholism and drug abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese outpatients with type 2 diabetes in Nanjing First Hospital who meet the the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Day 1
  Blood glycated hemoglobin
MBG | Day 1 to Day 4
  24 h mean blood glucose
MAGE | Day 1 to Day 4
  24 h mean amplitude of glycemic excursions
SDBG | Day 1 to Day 4
  the standard deviation of the MBG

CONTACTS AND LOCATIONS:
Overall Officials: Ma Jianhua, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hostital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wang H, Zhou Y, Wang Y, Cai T, Hu Y, Jing T, Ding B, Su X, Li H, Ma J. Basal Insulin Reduces Glucose Variability and Hypoglycaemia Compared to Premixed Insulin in Type 2 Diabetes Patients: A Study Based on Continuous Glucose Monitoring Systems. Front Endocrinol (Lausanne). 2022 Apr 27;13:791439. doi: 10.3389/fendo.2022.791439. eCollection 2022. PMID 35574003